CLINICAL TRIAL: NCT03664570
Title: ANTERO-3: The Impact of Enteral Nutrition Infusion Rate on Gastric Motility and Gastric Emptying Rate, Measured With the VIPUN Balloon Catheter, Magnetic Resonance Imaging and the 13C-octanoate Breath Test.
Brief Title: Enteral Nutrition Infusion Rate and Gastric Function
Acronym: ANTERO-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Dr Jan Tack (Other)
Responsible Party: Sponsor-Investigator, Prof Dr Jan Tack, Head of Clinic - Gastroenterology / Professor of Medicine / Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: S61853
Record Dates: First submitted 2018-08-29; First posted 2018-09-10 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: Gastric motility

STUDY DESIGN:
Intervention Model Description: Three-way crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Condition A (Experimental): * Infusion rate = 25 ml/h
  * Radiography: confirmation balloon position
  * VIPUN Balloon Catheter
  * 13C-Octanoate Breath Test o
  Interventions: Device: VIPUN Balloon Catheter
- Condition B (Experimental): * Infusion rate = 75 ml/h
  * Magnetic resonance imaging
  * VIPUN Balloon Catheter
  * 13C-Octanoate Breath Test
  Interventions: Device: VIPUN Balloon Catheter
- Condition C (Experimental): * Infusion rate = 250 ml/h
  * Magnetic resonance imaging
  * VIPUN Balloon Catheter
  * 13C-Octanoate Breath Testt
  Interventions: Device: VIPUN Balloon Catheter

INTERVENTIONS:
Device: VIPUN Balloon Catheter — The VIPUN Balloon Catheter is a nasogastric balloon catheter consisting of a standard nasogastric double lumen Sump catheter and a balloon attached to this catheter. Once the catheter is advanced into the stomach, the balloon can be inflated. The inflated balloon dimensions and intraballoon pressure are such that intragastric motility can optimally be assessed without inducing epigastric symptoms.
  Other Names: VIPUN system

SUMMARY:
A complex neurohumoral feedback mechanism regulates gastric emptying of enteral nutrition through changes in gastric motility. In this investigation, we aim to investigate the impact of different infusion rates of enteral nutrition on gastric motility, gastric emptying rate, epigastric symptoms and satiation.

Additionally, magnetic resonance imaging will be used to validate an extended 13C-octanoate breath test for gastric emptying of a liquid test meal that is infused over 2 hours. Furthermore, the reliability of a manual position check of the VIPUN Balloon catheter will be confirmed with radiographic imaging. Finally, the data will be used for the data driven optimization of the VIPUN MI algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* At least 18 years old
* BMI between and including 18 and 30
* Understand and able to read Dutch
* In good health on the basis of medical history
* Female subjects of childbearing potential are willing to use adequate contraception
* Refrains from herbal, vitamin and other dietary supplements on the day of the visits

Exclusion Criteria:

* Dyspeptic symptoms (assessed with PAGI-SYM questionnaire)
* Using any medication that might affect gastric function or visceral sensitivity
* Known / suspected current use of illicit drugs
* Known psychiatric or neurological illness
* Any gastrointestinal surgery that could influence normal gastric function in the opinion of the investigator
* History of heart or vascular diseases like irregular heartbeats, angina or heart attack
* Nasopharyngeal surgery in the last 30 days
* History of thermal or chemical injury to upper respiratory tract or esophagus
* Current esophageal or nasopharyngeal obstruction
* Known coagulopathy
* Known esophageal varices
* Metal or other MRI incompatible implants
* Contra-indications for MR (checked by MR safety questionnaire)
* Pregnancy
* Claustrophobia
* Have a known allergy or intolerance to cow milk, soy, saccharose or any other ingredient of Isosource Standard.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Motility | 8 hour
  Motility index (MI) measured with the VIPUN Balloon Catheter.
Gastric emptying rate (13C-Octanoate Breath Test) | 8 hour
  Gastric emptying rate of liquid test meal, measured with 13C-Octanoate Breath Test.
Gastric emptying rate (Magnetic resonance imaging) | Conditions B and C: 4 hour.
  Gastric emptying rate of liquid test meal, measured with magnetic resonance imaging

SECONDARY OUTCOMES:
Satiation | 6 hour
  Subjective satiation score at a 30-minute interval. Visual Analogue Scale (100 mm, 0=absent, 100= maximal sensation).
Safety profile VIPUN Balloon Catheter | Trough study completion, from Visit 1 until completion of Visit 3, on average 3 weeks
  Incidence, frequency, severity, seriousness and relatedness of AE's
Feasibility VIPUN Balloon Catheter related procedures | Trough study completion, from Visit 1 until completion of Visit 3, on average 3 weeks
  Success rate of completing the procedure (placement and removal VIPUN Balloon Catheter
Reliability manual position check | Once for each subject (during Condition A only): Position of the inflated balloon is judged on the thorax Rx (t<0) prior to start motility recording (= reference time point, t=0).
  Success rate (pass/fail) (reliability) of the manual position check of the VIPUN balloon catheter
Position catheter at t=480. | During Condition A only: at t=480 minutes (after cessation motility recording).
  Qualitative assessment of the migration of the catheter over the course of the study procedures.
Epigastric symptoms | 6 hours
  Subjective epigastric symptom scores at a 30-minute interval. 3 Visual Analogue Scales (100 mm, 0=absent, 100= maximal sensation). Scale 1: Nausea, Scale 2: Bloating, Scale 3: Pain.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No